CLINICAL TRIAL: NCT07316426
Title: Preoptimisation in Ventral Hernia Surgery- a Randomised Trial
Brief Title: Preoptimisation in Ventral Hernia Surgery
Acronym: PreOpt
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Region Norrbotten (Unknown); Region Västerbotten (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PreOpt
Record Dates: First submitted 2025-12-01; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-09

CONDITIONS: Hernia; Hernia, Ventral; Hernia Incisional; Hernia, Umbilical
Keywords: preoptimisation; prehabilitation
MeSH Terms: conditions — Hernia; Hernia, Ventral; Incisional Hernia; Hernia, Umbilical

STUDY DESIGN:
Intervention Model Description: This study is a prospective, single-blinded, multicentre, randomised, controlled superiority trial employing a parallel-group design with an allocation ratio of 1:1.
Who Masked: Outcomes Assessor
Masking Description: The surgeon responsible for the follow-up assessments at 3 and 12 months postoperatively will be blinded to the participant's allocation to either the intervention or the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group participates in a home-based, multimodal prehabilitation programme addressing physical inactivity, obesity, inadequate management of comorbidities, smoking, and alcohol consumption.
  Interventions: Procedure: preoptimisation programme
- control (No Intervention): The control group will receive basic guidance on physical activity and weight management during the preoperative consultation.

INTERVENTIONS:
Procedure: preoptimisation programme — The intervention group follows a home-based, multimodal prehabilitation programme targeting physical inactivity, obesity, comorbidities, smoking, and alcohol use. Designed to suit both rural and urban populations in northern Sweden, the programme lasts for a minimum of three months before surgery.
  Arms: Intervention

SUMMARY:
The study is a multicentre, single-blinded, randomised controlled trial. Ventral hernia patients with an aperture width between four and eight centimetres are randomised to either participation in a multimodal preoptimisation programme, including interventions to increase physical activity, promote weight loss, and optimise the treatment of comorbidities, or to surgery without structured preoptimisation. The primary endpoint is complications at three months postoperatively. During surgery, biopsies of skin, muscle, and fascia will be collected, along with pre- and postoperative blood samples, to analyse the molecular effects of preoptimisation, particularly in relation to collagen metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a ventral hernia with a defect width of at least 4 cm.
* Symptom burden related to the hernia sufficient to justify surgical intervention.
* Age ≥ 18 years.

Exclusion Criteria:

* Expected survival of less than three years.
* Inability to comprehend oral and written information or to provide informed consent.
* Acute complication of the hernia requiring emergency surgical intervention.
* General condition characterised by severe limitations in physical functional capacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Complications at three months postoperatively | 3 months postoperatively
  Incidence of surgical and medical (including anaesthetic) complications at 3 months postoperatively.

SECONDARY OUTCOMES:
Complications at twelve months postoperatively | 12 months postoperatively
  Incidence of surgical and medical complications at 12 months postoperatively.
Patient-reported pain | Measured at inclusion, preoperatively, 3 and 12 months postoperatively.
  Patient-reported pain measured with Ventral Hernia Pain Questionnaire, VHPQ. Max score is 40 and minimum score is 0, a lower score indicates less abdominal wall pain.
Quality of life with EQ-5D | Measured at inclusion, preoperatively, 3 and 12 months postoperatively.
  Quality of life assessed using the EuroQol 5-Dimensions questionnaire (EQ-5D index score). Max score is 1.0, which equals to perfect health and a lower score indicates lower quality of life with 0 is equivalent to death. Negative scores indicated health states considered worse than dead (e.g. severe disability).
Aesthetic outcome | Measured at clinical follow-upat 3 and 12 months postoperatively.
  Patient reported aestethic outcome measured with a Numerical Ratin Scale, NRS scale, range 1-10 where a higher score indicates better patient reported aesthetic outcome.
Recurrence rate | Measured at clinical follow-up at 3 and 12 months postoperatively.
  Recurrence of ventral hernia.
Change in physical activity | meassured close to inclusion and within a few weeks preoperatively.
  changes in physical activity measured with accelerometer for one week.
Weight | Measured at inclusion, preoperatively, 3 and 12 months postoperatively.
  Weight measured i kg.
Collagen metabolism | Biopsies will be taken perioperatively and thus be avalable for analysis when all study subjects have undergone surgery.
  Difference between study groups in the expression levels of a panel of markers of collagen degradation and synthesis (including CHP, Collagen 1 and 4, MMP) in tissue samples taken from fascia, muscle and skin.
Hba1c | at baseline, perioperatively, postoperative day 1, at follow up 3 and 12 months postoperatively.
  Hba1c in bloodsamples
Hernia aperature width | measured peroperatively and on preoperative ct-scan preinclusion or within a few weeks after inclusion
  Hernia aperature width
B-PETH | at baseline, perioperatively and at follow up at 3 and 12 months postoperatively.
  B-PETH
Rutine labarotory tests | At baseline, perioperatively, postoperative day 1, at follow up 3 and 12 months postoperatively
  Number of participants with abnormal routine laboratory tests results
Hyaluronan metabolism | Biopsies will be taken perioperatively and thus be avalable for analysis when all study subjects have undergone surgery.
  Difference between study groups in the expression patterns and histological distribution of hyaluronan and hyaluronan metabolism-related factors (including CD44, TRAMM, and hyaluronidases) in tissue samples taken from fascia, muscle and skin.

CONTACTS AND LOCATIONS:
Locations (5):
- Sweden (5):
  - Gällivare hospital, Gällivare, Norrbotten County
  - Sunderby Hospital, Luleå, Norrbotten County
  - Lycksele Hospital, Lycksele, Västerbotten County
  - Skellefteå Hospital, Skellefteå, Västerbotten County
  - Umeå University Hospital, Umeå, Västerbotten County

IPD SHARING:
Plan to Share IPD: No